CLINICAL TRIAL: NCT07240623
Title: A Randomized Controlled Single-blind Clinical Trial Comparing the Therapeutic Effects of Manual Acupuncture at Distal Acupoints With Electroacupuncture at Local Acupoints in Patients With Acute Neck Pain Due to Cervical Spondylosis
Brief Title: Comparison of Manual Acupuncture at Distal Acupoints Versus Electroacupuncture at Local Acupoints in Patients With Acute Neck Pain Due to Cervical Spondylosis
Acronym: DALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Medicine - Vietnam National University at Ho Chi Minh city (Other)
Responsible Party: Principal Investigator, Nguyen Ky Xuan Nhi, Medical Specialist, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3836/QĐ-ĐHYD; IRB No. IRB-VN01002 (Other: Approved by the Institutional Review Board of University of Medicine and Pharmacy at Ho Chi Minh)
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cervical Spondylosis; Acute Neck Pain; Neck Pain Musculoskeletal; Degenerative Cervical Spine
MeSH Terms: conditions — Spondylosis | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Acupuncture (Active Comparator): Participants receive manual acupuncture at distal acupoints (SI3, SI5, TE4, BL60, BL62, GB40) on the contralateral side of the painful neck area for 25 minutes. During needle retention, patients perform active cervical spine movements (flexion, extension, lateral flexion, and rotation) for at least 10 minutes.
  Interventions: Procedure: Manual acupuncture at distal acupoints
- Electroacupuncture (Active Comparator): Participants receive electroacupuncture for 25 minutes at local acupoints (GB20-SI15 and GB21-LU7) on the painful side. After needle removal, patients perform active cervical spine movements (flexion, extension, lateral flexion, and rotation) for at least 10 minutes.
  Interventions: Procedure: Electroacupuncture at local acupoints

INTERVENTIONS:
Procedure: Manual acupuncture at distal acupoints — Manual acupuncture applied for 25 minutes at distal acupoints selected based on meridian diagnosis (SI3, SI5, TE4, BL60, BL62, GB40) on the contralateral side of the pain. During needle retention, participants performed active cervical spine movements (flexion, extension, lateral flexion, and rotation) for at least 10 minutes.
  Other Names: Manual acupuncture; Distal acupoints
  Arms: Manual Acupuncture
Procedure: Electroacupuncture at local acupoints — Electroacupuncture applied for 25 minutes at local acupoints (GB20-SI15 and GB21-LU7) on the painful side. After needle removal, participants performed active cervical spine movements (flexion, extension, lateral flexion, and rotation) for at least 10 minutes.
  Other Names: Electroacupuncture; Local acupoints
  Arms: Electroacupuncture

SUMMARY:
This study is a randomized, single-blind, controlled clinical trial involving two groups: manual acupuncture and electroacupuncture, with 62 participants in each group. All participants received treatment once daily for 10 consecutive days, combined with at least 10 minutes of active cervical spine exercises per session.

Participants were allowed to take one 500 mg tablet of paracetamol if the pain exceeded their tolerance threshold, with a minimum interval of 6 hours between doses and a maximum daily dose of 1,500 mg. The number of tablets taken each day was recorded. No other analgesic interventions were permitted during the study period.

The objective of this study was to compare and evaluate the effectiveness of the two interventions in improving pain intensity (VAS score) and limitations of cervical range of motion after each treatment session. In addition, adverse events were monitored and recorded after every intervention.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of neck pain lasting less than 6 weeks.
* Pain intensity ≥ 50 mm on the Visual Analogue Scale (VAS).
* Presence of limitation in at least one cervical range of motion (ROM).
* Radiographic diagnosis of cervical spondylosis based on Kellgren and Lawrence criteria.

Exclusion Criteria:

* Patients with infection, cachexia, or psychiatric disorders.
* Currently using analgesic medication.
* Cervical movement limitation persisting for more than 6 weeks.
* History of or indication for cervical spine surgery.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity (VAS score) | Baseline and after each daily treatment for 10 consecutive days
  Pain intensity is assessed using a 100 mm Visual Analogue Scale (VAS), where ≤4 indicates no pain and 100 indicates the worst imaginable pain. The change in VAS score from baseline to each treatment day is recorded for comparison between groups.
Change in cervical range of motion (ROM) limitation score | Baseline and after each daily treatment for 10 consecutive days
  The cervical range of motion (ROM) was measured for six movements: flexion, extension, right and left lateral flexion, and right and left rotation. Each movement was assessed using a goniometer, and the measured angles were converted into a limitation score ranging from 0 to 4 according to the following grading system:
  * 0 - Normal ROM (flexion 45°-55°, extension 60°-70°, lateral flexion 40°-50°, rotation 60°-70°)
  * 1 - Mild limitation (flexion 40°-44°, extension 55°-59°, lateral flexion 35°-39°, rotation 55°-59°)
  * 2 - Moderate limitation (flexion 35°-39°, extension 50°-54°, lateral flexion 30°-34°, rotation 50°-54°)
  * 3 - Severe limitation (flexion 30°-34°, extension 45°-49°, lateral flexion 25°-29°, rotation 45°-49°)
  * 4 - Very severe limitation (<30° flexion, <45° extension, <25° lateral flexion, <45° rotation) The total limitation score was calculated as the sum of all six movement scores, with higher scores indicating greater cervical movement restriction.

SECONDARY OUTCOMES:
Adverse events related to acupuncture or electroacupuncture | Monitored immediately after each treatment session and at the end of the 10-day treatment period
  Any adverse events such as local pain, swelling, dizziness, or fainting were observed and recorded after each treatment session. Severity and frequency were summarized descriptively.

OTHER OUTCOMES:
Number of paracetamol tablets used | Recorded daily during the 10-day treatment period
  Participants were allowed to take one 500 mg tablet of paracetamol at ≥6-hour intervals if the pain exceeded their tolerance, with a maximum dose of 1500 mg/day. The number of tablets used per day was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Traditional Medicine Hospital of Ho Chi Minh City, Ho Chi Minh City, Xuan Hoa Ward, Vietnam

IPD SHARING:
Plan to Share IPD: No